CLINICAL TRIAL: NCT06898151
Title: Carotid Endarterectomy and Stenting Timing：The CEST Trial
Brief Title: Carotid Endarterectomy and Stenting Timing
Acronym: CEST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEST
Record Dates: First submitted 2025-03-03; First posted 2025-03-27 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Carotid Endarterectomy; Carotid Stenting
Keywords: Timing of carotid artery revascularization

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CEA/CAS within 48 hours after randomization (Experimental): All the participants in this group will be performed with CEA/CAS plus best medical treatment including Aspirin 100mg per day + Clopidogrel 75mg per day or Ticagrelor 90mg twice per day before surgery. If CEA was assigned, mono anti-platelet therapy will be performed thereafter. If CAS was assigned, dual-antiplatelet will be performed for 3 months after surgery followed by mono anti-platelet therapy thereafter. CAS or CAS will be performed within 48h after randomization.
  Interventions: Procedure: CEA/CAS plus best medical treatment
- CEA/CAS after 14 days of randomization (Other): All the participants in this group will be performed with CEA/CAS plus best medical treatment including Aspirin 100mg per day + Clopidogrel 75mg per day or Ticagrelor 90mg twice per day before surgery. If CEA was assigned, mono anti-platelet therapy will be performed thereafter. If CAS was assigned, dual-antiplatelet will be performed for 3 months after surgery followed by mono anti-platelet therapy thereafter. CEA or CAS will be performed 14 days after randomization.
  Interventions: Procedure: CEA/CAS plus best medical treatment

INTERVENTIONS:
Procedure: CEA/CAS plus best medical treatment — Timing of CEA/CAS plus best medical treatment

SUMMARY:
To compare the safety and efficacy of carotid revascularization performed within 48 hours versus after 14 days in patients with symptomatic carotid stenosis accompanied with MRI-confirmed acute infarction (high signal on diffusion-weighted imaging accompanied by low apparent diffusion coefficient signal) in the responsible vascular territory.

DETAILED DESCRIPTION:
Carotid artery stenosis is an important cause of stroke, and about 20-30% of ischemic stroke can be attributed to carotid artery stenosis. In the past 20 years, the prevalence of carotid artery stenosis in my country has increased by 70.07%, which has imposed a heavy burden on the national economy and society. At present, for symptomatic carotid artery stenosis, carotid artery revascularization, mainly carotid endarterectomy (CEA) and carotid artery stenting (CAS), combined with optimal drug therapy (antiplatelet + lipid-lowering), has become the mainstream treatment. In 2004, Rothwell et al. conducted a meta-analysis of individual case data from the European Carotid Surgery Trial (ECST) and the North American Symptomatic Carotid Endarterectomy Trial (NASCET). The results showed that when the waiting time between the onset of symptoms and the receipt of revascularization was prolonged, the effect of carotid artery revascularization in preventing future strokes would be significantly weakened. The latest guidelines issued by the European Stroke Organisation (ESO) recommend that 50-99% of patients with symptomatic carotid stenosis undergo acute CEA, preferably within 14 days after the ischemic event. Based on these clinical research evidence, an increasing number of patients have undergone acute CEA over the past two decades. For example, a study in the United States confirmed that the median waiting time from the occurrence of an ischemic event to receiving CEA decreased from 22 days in 2009 to 12 days in 2014, and the proportion of patients treated within the 14-day interval increased from 37% to 58%. Similarly, data from Germany from 2003 to 2014 showed that the interval from the ischemic event to receiving CEA decreased from 28 days to 8 days. Despite this, in China, the proportion of patients who received carotid revascularization within 14 days is still relatively low due to concerns about increased perioperative complications of acute revascularization.

Previously, the investigators retrospectively analyzed 1172 patients with symptomatic carotid stenosis, and used diffusion-weighted imaging (DWI) and apparent diffusion coefficient (ADC) sequences to identify whether there was acute new infarction before surgery. Further analysis found that for patients with symptomatic carotid stenosis combined with acute new infarction, regardless of the type of revascularization (CEA or CAS), the risk of postoperative serious adverse events was significantly increased. Therefore, for patients with preoperative new infarction on MRI, the investigators urgently need more effective treatment strategies to reduce the incidence of postoperative adverse events and improve the long-term prognosis of patients. The discussion of the timing of surgery is an important part of the treatment strategy. However, there is no large-scale clinical study report on whether preoperative new infarction on MRI has an auxiliary effect on the optimal timing of surgery for symptomatic carotid artery stenosis. Therefore, the investigators plan to initiate a multicenter, prospective, randomized, open-label, blinded RCT trial to explore whether preoperative new infarction on MRI can serve as a new marker for the safety and effectiveness of revascularization surgery in patients with symptomatic carotid artery stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Diagnosed with symptomatic carotid stenosis, defined as the occurrence of sudden-onset neurological symptoms within the territory of the responsible artery within 180 days before randomization (e.g., contralateral hemiparesis, slurred speech/difficulty in expression, ipsilateral monocular vision loss, etc.);
* Stenosis located in the extracranial segment of the internal carotid artery (with or without involvement of the adjacent common carotid artery);
* Degree of stenosis in the responsible carotid artery confirmed to be ≥50% and ≤99% by CTA/MRA/DSA, based on NASCET criteria;
* Brain MRI within 72 hours before randomization indicating an acute infarction in the responsible vascular territory, characterized by high signal on DWI and low signal on ADC;
* Modified Rankin Scale (mRS) score <3;
* Written informed consent obtained from the patient or their legal representative.

Exclusion Criteria:

* Progressive neurological deterioration within 72 hours before randomization, defined as an increase in mRS score by ≥2 points or NIHSS score by ≥4 points;
* Brain MRI within 72 hours before randomization indicating a large infarction (infarct size > 1/2 of the middle cerebral artery territory);
* MRI evidence of hemorrhagic cerebrovascular diseases (e.g., brain tumor, brain abscess, vascular malformations) or other non-ischemic cerebrovascular diseases (e.g., multiple sclerosis);
* Non-atherosclerotic carotid stenosis (e.g., carotid artery dissection, carotid web, floating thrombus, fibromuscular dysplasia, Takayasu arteritis, etc.);
* Need for simultaneous surgical intervention for tandem lesions in the ipsilateral carotid artery or other vascular surgeries;
* History of cerebrovascular surgery within 6 months before randomization;
* Coexisting cerebrovascular stenosis requiring revascularization within 3 months after randomization;
* History of spontaneous intracranial hemorrhage within 12 months before randomization;
* Clear indication for anticoagulation therapy (suspected cardiac embolic source such as atrial fibrillation, known mechanical heart valve, or suspected infective endocarditis);
* Laboratory abnormalities, including white blood cell count < 2×10⁹/L, hematocrit < 30%, platelet count < 100×10⁹/L, INR > 1.5, or heparin-induced thrombocytopenia;
* Inability to use antiplatelet therapy due to specific reasons, such as active gastrointestinal ulcers, gastrointestinal bleeding within the past 3 months, known severe allergy, severe renal insufficiency (creatinine >1.5 times the normal upper limit), hepatic dysfunction (ALT or AST >2 times the normal upper limit), or severe heart failure (NYHA Class III-IV);
* Presence of other severe diseases that may affect adherence to the study protocol, such as severe infection, advanced chronic obstructive pulmonary disease (COPD), active malignant tumors, dementia, psychiatric disorders, or uncontrolled severe hypertension;
* Pregnant or breastfeeding women who are not in menopause;
* Participation in another investigational device or drug trial that may interfere with this study;
* Any other medical condition or history that, in the investigator's judgment, may affect the efficacy or safety assessment of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2025-03-07 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Any stroke, death, myocardial infarction, or urgent revascularization from randomization to 30 days, or an ischemic stroke in the responsible vascular territory occurring between 30 days and 3 months post-randomization. | From randomization to 3 months
  Urgent revascularization indicates the rescue surgery when transient ischemic attack happened during medical treatment. TIA: any temporary neurological deficit lasting less than 24 hours confirmed by a certified neurologist. Stroke including ischemic and hemorrhagic stroke within the territory of the treated carotid artery as confirmed by cerebral MRI or CT. All cause death will be confirmed when mRS scale is 6. Myocardial infarction: detection of rise and/or fall of cardiac biomarkers with at least one value above the 99th percentile of the upper reference limit together with evidence of myocardial ischaemia with at least one of the following: symptoms of ischaemia, ECG changes indicative of new ischaemia (new ST-T changes or new left bundle branch block, new onset of pathological Q waves in ECG, imaging evidence of new loss of viable myocardium or new regional wall motion abnormolity.

SECONDARY OUTCOMES:
Ischemic stroke in the responsible vascular territory | 30 days and 3 months post-randomization
  The ischemic stroke will be confirmed when infarction of responsible vascular territory could be identified on cerebral MRI or CT.
Any stroke | from randomization to 3 months post-randomization
  The ischemic or hemorrhagic stroke will be confirmed by cerebral MRI or CT.
Disabling stroke (mRS>3) | from randomization to 3 months
  The modified Rankin Scale (mRS) will be used to define this outcome. The disabling stroke is confirmed when mRS>3. The mRS is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. It has become the most widely used clinical outcome measure for stroke clinical trials.
Fatal stroke | from randomization to 3months
  Ischemic or hemorrhagic stroke (confirmed on cerebral MRI) leading to death.
Hemorrhagic stroke | from randomization to 3 months
  The hemorrhagic stroke need to be confirmed by cerebral MRI or CT
Death | from randomization to 3 months
  All cause of death as confirmed by mRS=6.
Any stroke, death, myocardial infarction | from randomization to 3 months
  Stroke: Including ischemic and hemorrhagic stroke as confirmed by cerebral CT or MRI.
  Death: All cause of death as confirmed by mRS=6. Myocardial infarction: detection of rise and/or fall of cardiac biomarkers (preferable troponin) with at least one value above the 99th percentile of the upper reference limit together with evidence of myocardial ischemia with at least one of the following: symptoms of ischemia, ECG changes indicative of new ischemia (new ST-T changes or new left bundle branch block, new onset of pathological Q waves in ECG, imaging evidence of new loss of viable myocardium or new regional wall motion abnormality).
Myocardial infarction | from randomization to 3 months
  Myocardial infarction: detection of rise and/or fall of cardiac biomarkers (preferable troponin) with at least one value above the 99th percentile of the upper reference limit together with evidence of myocardial ischemia with at least one of the following: symptoms of ischemia, ECG changes indicative of new ischemia (new ST-T changes or new left bundle branch block, new onset of pathological Q waves in ECG, imaging evidence of new loss of viable myocardium or new regional wall motion abnormality)
Proportional distribution of mRS/NIHSS | 3 months post-randomization
  The mRS score range from 0 (no disability) to 6 (death); the NIHSS score range from 0 (no disability) to 42 (severely disabled).
EQ-5D-5L | 3 months post-randomization
  The EQ-5D 5-Levels (EQ-5D-5L) range from 5 (no problems) to 25 (extreme problems), which deceased patients have a utility of 0.
Rehospitalization | from randomization to 3 months
  Times of rehospitalization.
Ischemic stroke or urgent revascularization | Randomization to surgery
  Ischemic stroke will be confirmed by cerebral CT or MRI. Urgent revascularization indicated to those who suffered from transient ischemic stroke (TIA) and received urgent surgery. TIA: any temporary neurological deficit lasting less than 24 hours confirmed by a certified neurologist.
Any stroke, death and myocardial infarction | surgery to 30 days
  Stroke: Including ischemic and hemorrhagic stroke as confirmed by cerebral CT or MRI. Death: All cause of death as confirmed by mRS=6. Myocardial infarction: detection of rise and/or fall of cardiac biomarkers (preferable troponin) with at least one value above the 99th percentile of the upper reference limit together with evidence of myocardial ischemia with at least one of the following: symptoms of ischemia, ECG changes indicative of new ischemia (new ST-T changes or new left bundle branch block, new onset of pathological Q waves in ECG, imaging evidence of new loss of viable myocardium or new regional wall motion abnormality).
Average hospital stay | from randomization to 3 months
  The average days of hospital stay will be recorded and the proportion will be presented.
Average hospital cost | from randomization to 3 months
  The average cost before reimbursement will be recorded and the proportion will be presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University., Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Naylor R, Rantner B, Ancetti S, de Borst GJ, De Carlo M, Halliday A, Kakkos SK, Markus HS, McCabe DJH, Sillesen H, van den Berg JC, Vega de Ceniga M, Venermo MA, Vermassen FEG, Esvs Guidelines Committee, Antoniou GA, Bastos Goncalves F, Bjorck M, Chakfe N, Coscas R, Dias NV, Dick F, Hinchliffe RJ, Kolh P, Koncar IB, Lindholt JS, Mees BME, Resch TA, Trimarchi S, Tulamo R, Twine CP, Wanhainen A, Document Reviewers, Bellmunt-Montoya S, Bulbulia R, Darling RC 3rd, Eckstein HH, Giannoukas A, Koelemay MJW, Lindstrom D, Schermerhorn M, Stone DH. Editor's Choice - European Society for Vascular Surgery (ESVS) 2023 Clinical Practice Guidelines on the Management of Atherosclerotic Carotid and Vertebral Artery Disease. Eur J Vasc Endovasc Surg. 2023 Jan;65(1):7-111. doi: 10.1016/j.ejvs.2022.04.011. Epub 2022 May 20. No abstract available. PMID 35598721
- [Background] Rothwell PM, Eliasziw M, Gutnikov SA, Warlow CP, Barnett HJ; Carotid Endarterectomy Trialists Collaboration. Endarterectomy for symptomatic carotid stenosis in relation to clinical subgroups and timing of surgery. Lancet. 2004 Mar 20;363(9413):915-24. doi: 10.1016/S0140-6736(04)15785-1. PMID 15043958